CLINICAL TRIAL: NCT05632393
Title: A Prospective, Open-label, Single-dose Phase 1 Study to Measure Daridorexant in Breast Milk of Healthy Lactating Women
Brief Title: A Study to Measure Daridorexant in Breast Milk of Healthy Lactating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-078-122
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daridorexant 50 mg (Experimental): Daridorexant 50 mg will be administered once in the morning of Day 1.
  Interventions: Drug: Daridorexant

INTERVENTIONS:
Drug: Daridorexant — Daridorexant will be available as film-coated tablets for oral administration formulated at a strength of 50 mg.

SUMMARY:
A study to measure daridorexant in breast milk of healthy lactating women

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy lactating female subject aged at least 18 years at Screening.
* Female subject who has delivered a term infant (≥ 37 weeks' gestation) and who is breastfeeding her infant (and/or pumping) for at least 2 weeks postpartum at Screening; lactation must be well-established to maintain an adequate milk supply with regular breastfeeding (and/or pumping, e.g., 3 to 4 times per day and not providing more than 1 supplemental bottle of formula per day and the infant has not started eating solids). Subjects planning on weaning their infants after enrollment who meet the afore mentioned requirements will be considered for enrollment in the study.
* Agreement to refrain from breastfeeding any infant with her own milk from Day -1 up to 72 h after study treatment administration.
* Ability of subject's infant to feed from a bottle or no anticipated compromise of subject's infant's nutrition with time period of refraining from breastfeeding planned during the study.
* Agreement to collect breast milk from pre-dose (directly prior to study treatment administration) to Day 4 (72 h after study treatment administration) using an electric pump provided by the study site.
* Must agree to use an acceptable effective method of contraception consistently and correctly (e.g., oral progestin-only contraceptive; implants; intra uterine devices; male or female condom with or without spermicide; cap, diaphragm or sponge with spermicide) from Screening up to at least 72 h after study treatment administration, be sexually inactive, or be in same-sex relationship.

Exclusion Criteria:

* Known hypersensitivity to daridorexant or treatments of the same class, or any of its excipients.
* History of narcolepsy.
* Mastitis or other condition that prevents the collection of breast milk from one or both breasts at Screening or on Day -1.
* History of breast implants, breast augmentation, or breast reduction surgery which prevents the collection of breast milk.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Milk pharmacokinetic endpoints: Amount of daridorexant excreted (mg) | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
  Cumulative amount excreted in breast milk over the collection time

OTHER OUTCOMES:
Milk pharmacokinetic endpoints: Fraction (percentage) of dose excreted in breast milk | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
Milk pharmacokinetic endpoints: Relative infant daridorexant dose (percentage) | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
  Percentage of dose that would be consumed by the infant, adjusted to maternal weight and infant weight on Day -1
Plasma pharmacokinetic endpoints: Cmax | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
Plasma pharmacokinetic endpoints: Tmax | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
Plasma pharmacokinetic endpoints: AUC0-inf | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
Plasma pharmacokinetic endpoints: T1/2 | 0 to 72 hours after study treatment administration (Total duration: up to 4 days)
Treatment-emergent (S)AEs | Up to end of study (EOS; total duration: up to 46 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idosia Pharmaceuticals Ltd
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No